CLINICAL TRIAL: NCT02834455
Title: Rational Approach to Unilateral Pleural Effusion in Patients Suspected of Malignancy. Efficacy, Pain, Quality of Life, and Economy
Brief Title: Rational Approach to a Unilateral Pleural Effusion2
Acronym: REPEAT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Patient inclusion cannot be reached within timelimits
Sponsor: Simon Reuter (Other)
Responsible Party: Sponsor-Investigator, Simon Reuter, MD, Naestved Hospital
Organization: Naestved Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Resp-REPEAT-SIRE
Record Dates: First submitted 2015-06-17; First posted 2016-07-15 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Lung Neoplasms
Keywords: Thoracoscopy
MeSH Terms: conditions — Lung Neoplasms | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CE-CT scanning (Active Comparator): Contrast-enhanced CT scan of the thorax and abdomen.
  Interventions: Device: Contrast-enhanced CT
- PET-CT scanning (Active Comparator): Positron-emission-CT scanning (low dose without contrast) of the thorax and abdomen.
  Interventions: Device: PET-CT

INTERVENTIONS:
Device: Contrast-enhanced CT — 50% of patients with unilateral pleural effusion will have performed a CE-CT
  Arms: CE-CT scanning
Device: PET-CT — 50% of patients with unilateral pleural effusion will have performed a PET-CT
  Arms: PET-CT scanning

SUMMARY:
Recurrent unilateral, non-infectious pleural exudate is suspicious for primary or secondary pleural malignancy. Both conditions are associated with 5-year survival of 10%. Work-up is difficult, as the pleural surface is large and <33% of pleural malignancies shed malignant cells to the pleural fluid. Even so, additional tissue biopsies are needed for establishing mutation status for targeted therapies.

Optimal imaging to guide tissue sampling is pivotal. PET-CT has higher sensitivity than conventional CT for detecting malignant lesions >10mm. However, no randomised trial has investigated differences in diagnostic accuracy, time-to-diagnosis, or economics. Falsely PET-positive lesions in e.g. colon however, lead to more derived tests than do CT alone.

Gold standard for pleural tissue sampling is the surgical (VATS) thoracoscopy, allowing direct visual guiding of tissue sampling from all pleural surfaces. Yet, globally the medical (pleuroscopy) thoracoscopy is more widely used: cheaper, outpatient procedure, but allows only sampling from the parietal pleura. To date, no randomised studies have compared medical and surgical thoracoscopy concerning diagnostic hit rates, adverse events, or economics.

The investigators will perform two randomized studies to investigate whether

1. PET/CT is comparable to CT alone
2. VATS is comparable to pleuroscopy concerning hit rate, total investigations performed, time-to-diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with recurrent pleural effusion of unknown origin after a first pleural tap according to BTS guidelines.
2. Indication for thoracoscopy according to BTS guidelines.
3. Patients accept further investigation according to Danish and BTS guidelines.
4. Have received oral and written consent and agreed.
5. At the time of inclusion, above 18 years of age.

Exclusion Criteria:

1. Female patients: pregnancy or breastfeeding.
2. Lack of language comprehension.
3. Legally incompetent patients.
4. Life expectancy less than 3 month.
5. Contraindications to pleural tissue sampling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Number of diagnostic thoracoscopies (either MT or VATS) | 2 years

SECONDARY OUTCOMES:
Number of derived investigations (i.e. gastroscopy, coloscopy) | 2 years
Number of patients diagnosed with cancer (cancer = an unequivocal diagnosis of neoplastic disease; no cancer = clinically benign cause, and improved imaging at 6 month control) | 2 years
Patient satisfaction and patient perceived discomfort | 2 years
  Using QLQC 30
Total costs calculated as costs patient-related, procedure-related, and overall | 2 years
Total procedures before cancer-diagnosis (cancer = yes/no) | 2 years
Patient satisfaction and patient perceived discomfort | 2 years
  EuroQol Q-5D a standardised instrument for use as a measure of health outcome

CONTACTS AND LOCATIONS:
Overall Officials: Uffe Boedtger, MD, PhD, Study Director — ubt@regionsjaelland.dk
Locations (1):
- Naestved Sygehus, Næstved, Denmark